CLINICAL TRIAL: NCT05096377
Title: The Effect of Erector Spinae Plane Block on Hemidiaphragm Paresis in Shoulder Surgery
Brief Title: Hemi-diaphragmatic Paresis and Erector Spinae Plane Block
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 8/12
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia, Regional; Shoulder
Keywords: Regional Anesthesia; Shoulder Surgery; Hemidiaphragmatic Paresis; Erector Spinae Plane Block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESP block group: Diaphragmatic excursion was measured using M-mode ultrasound during normal breathing, deep breathing and with the sniff manoeuvre.
  Interventions: Other: ESP block

INTERVENTIONS:
Other: ESP block — ESP block performed using ultrasound guidance. Diaphragmatic excursion was measured using M-mode ultrasound during normal breathing, deep breathing and with the sniff manoeuvre.

SUMMARY:
To assess the incidence of hemi-diaphragmatic paresis following ultrasound-guided erector spinae plane (ESP) block

DETAILED DESCRIPTION:
The aim of the study is to assess the effect of hemi-diaphragmatic paresis following ultrasound-guided erector spinae plane block.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 85 years
* American Society of Anesthesiology (ASA) I-III
* elective shoulder surgery

Exclusion Criteria:

* patient's refusal
* under 18 years of age or over 65 years of age
* ASA IV and above
* known allergy to local anaesthetic drugs
* the block cannot be applied due to bleeding disorders or localized skin infection at the injection site
* history of neurological and/or neuromucular disease
* history of severe bronchopulmonary disease
* a moderate to severe decrease in preoperative pulmonary function, or abnormality in preoperative chest radiography data (pleural effusion, pneumothorax, or hemidiaphragm elevation)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: shoulder surgery
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
incidence of hemi-diaphragmatic paresis | 30 minutes
  Diaphragmatic excursion was measured using M-mode ultrasound during normal breathing, deep breathing and with the sniff manoeuvre.

SECONDARY OUTCOMES:
intraoperative opioid consumption | 2 hour
  intraoperative opioid consumption will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, Principal Investigator — Antalya TRH; Ali Sait Kavaklı, Principal Investigator — Antalya TRH
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Muratpaşa, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Sivashanmugam T, Maurya I, Kumar N, Karmakar MK. Ipsilateral hemidiaphragmatic paresis after a supraclavicular and costoclavicular brachial plexus block: A randomised observer blinded study. Eur J Anaesthesiol. 2019 Oct;36(10):787-795. doi: 10.1097/EJA.0000000000001069. PMID 31397702